CLINICAL TRIAL: NCT07402876
Title: A Prospective, Randomized, Double-masked, Dosing-frequency-controlled, Multicenter Clinical Trial Evaluating the Safety and Activity of Intravitreally Injected ADX-2191 (Methotrexate Injection USP) in Patients With Primary Vitreoretinal Lymphoma
Brief Title: A Clinical Trial Evaluating Patients With Primary Vitreoretinal Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADX-2191-PVRL-001
Record Dates: First submitted 2026-01-29; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Primary Vitreoretinal Lymphoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Induction/Consolidation/Maintenance (ICM) ADX-2191 injection (Experimental)
  Interventions: Drug: ICM ADX-2191 injection
- Monthly ADX-2191 injection (Active Comparator)
  Interventions: Drug: Monthly ADX-2191 injection

INTERVENTIONS:
Drug: ICM ADX-2191 injection — Following the development of lymphomatous vitreous cells in at least one eye, subjects will follow ICM dosing with ADX-2191 intravitreal injections twice weekly for four weeks, followed by weekly for eight weeks, for a total of sixteen injections.
  Arms: Induction/Consolidation/Maintenance (ICM) ADX-2191 injection
Drug: Monthly ADX-2191 injection — Following the development of lymphomatous vitreous cells in at least one eye, subjects will dose monthly with ADX-2191 intravitreal injections for a total of three injections. Sham injections will be performed for those visits during which ADX-2191 is not injected, for a total of thirteen sham injections.
  Arms: Monthly ADX-2191 injection

SUMMARY:
A prospective, randomized, double-masked, dosing-frequency-controlled, multicenter clinical trial evaluating the safety and activity of intravitreally injected ADX-2191 (methotrexate injection USP) in patients with primary vitreoretinal lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. 21 years old or older; of any gender
2. Biopsy proven primary vitreoretinal lymphoma
3. Presence of lymphomatous vitreous cells at the Screening Visit and/or any eye that has been vitrectomized to confirm the diagnosis of primary vitreoretinal lymphoma
4. Willingness to participate in the clinical trial as evidenced by signing of an informed consent

Exclusion Criteria:

1. Known allergy or hypersensitivity to methotrexate
2. Planned eye surgery during the clinical trial
3. Women of childbearing potential who are pregnant or lactating
4. Pre-existing ocular or non-ocular conditions or diseases that, in the opinion of the investigator, could interfere with the conduct or interpretation of the clinical trial
5. Use of systemic methotrexate within one week prior to treatment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of clearance of lymphomatous vitreous cells compared across ICM and monthly ADX-2191 treatment groups after eight weeks of treatment | Eight weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Bascom Palmer Eye Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No